CLINICAL TRIAL: NCT02144363
Title: A Prospective Study of Diaphragmatic Electrical Activity in Preterm Infants as a Means to Predict Extubation Success
Brief Title: Electrical Activity of Diaphragm as a Means to Predict Extubation Success in Preterm Infants
Acronym: Edi
Status: Completed | Type: Observational
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Neetu Singh, Assistant Professor of Pediatrics, Dartmouth-Hitchcock Medical Center
Other Study IDs: D14057
Record Dates: First submitted 2014-04-30; First posted 2014-05-22 (Estimated); Last update posted 2016-03-11 (Estimated); Status verified 2016-03

CONDITIONS: Respiratory Distress Syndrome
Keywords: Preterm; RDS; Mechanical Ventilation; Extubation failure
MeSH Terms: conditions — Respiratory Distress Syndrome; Premature Birth

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Mechanical ventilation used to support the sick newborn infant is associated with many complications including the development of chronic lung disease. Limiting prolonged invasive ventilation remains an important strategy to decrease lung injury and prevent chronic lung disease. Currently, there is no objective measure available to predict readiness for removal of the endotracheal tube ("extubation") and discontinuing mechanical ventilation in this fragile population.

The investigators propose to predict extubation success by evaluating the electrical activity of the diaphragm (Edi), which provides important information about the "drive" to breathing coming from the brain and the function of the diaphragm, two essential factors determining extubation readiness and success.

DETAILED DESCRIPTION:
In this observational study, very low birth weight preterm infants with RDS who require mechanical ventilation in first 24 hour of life will be recruited. A size appropriate nasogastric tube with multiple array of electrodes (Edi catheter) will be inserted in each eligible infant. The average EdI (Edi_avg) will be measured during mechanical ventilation just before extubation. All infants will be extubated to non-invasive positive pressure ventilation (NIPPV or CPAP) delivered through nasal cannula

The specific aim is to determine whether there is a relationship between Edi_avg before extubation and the extubation success in a sample of preterm infants with respiratory distress syndrome (RDS). We hypothesize that Edi-avg of infants with successful extubation will be significantly different from the infants who fail extubation

ELIGIBILITY:
Inclusion Criteria:

Preterm infants less than 35 week gestation, requiring intubation and mechanical ventilation for respiratory distress in the first 24 hours of life

Exclusion Criteria:

Infants with a non-intact esophagus (e.g tracheal-esophageal fistula or atresia), a non-functional diaphragm (e.g. phrenic nerve palsy), severe intracranial hemorrhage or structural CNS abnormality, severe birth asphyxia and critically sick infant needing paralysis or deep sedation.

Ages: 1 Hour to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A convenience sample of forty(40) preterm infants less than 35 week gestation admitted in the ICN with the need for intubation and mechanical ventilation for respiratory distress in the first 24 hours of life will be recruited for this study.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Actual)
Dates: Start 2014-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Edi_avg just prior to extubation in infants with extubation success and those with extubation failure | From time of initial intubation to 3 days after extubation from mechanical ventilator
  Edi_avg prior to extubation will be compared between the group with successful extubation and those with failed extubation( i.e.needing re-intubation within 3 days of extubation)

SECONDARY OUTCOMES:
Study the trends of Edi_avg in preterm infants with respiratory distress syndrome requiring mechanical ventilation in first seven days of life. | First seven days of life
  Edi_avg will be recorded continuously during mechanical ventilation to a maximum of seven day. We hypothesize that Edi_avg would correlate with severity of respiratory distress ( measured by respiratory severity index, FiO2 X Mean airway pressure)

CONTACTS AND LOCATIONS:
Overall Officials: Neetu Singh, MD, MPH, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth Hitchcock Medcial Center, Lebanon, New Hampshire, United States

REFERENCES:
- [Derived] Singh N, McNally MJ, Darnall RA. Does Diaphragmatic Electrical Activity in Preterm Infants Predict Extubation Success? Respir Care. 2018 Feb;63(2):203-207. doi: 10.4187/respcare.05539. Epub 2017 Nov 28. PMID 29184049